CLINICAL TRIAL: NCT02383004
Title: Acupuncture for the Prevention of Emergence Delirium in Children Undergoing Myringotomy Tube Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Christine Martin, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00010770
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Delirium; Psychomotor Agitation
Keywords: myringotomy tubes; acupuncture; emergence delirium; pediatrics; general anesthesia
MeSH Terms: conditions — Delirium; Psychomotor Agitation; Emergence Delirium | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Same premedication, induction and maintenance protocol as the No Acupuncture (Standard of Care) group.
  The intervention will be placement of 4 acupuncture needles. The needles will be placed after inhalational anesthesia induction and removed prior to leaving the operating room. A total of 4 needles will be placed, one in each wrist at the HT7 point and one in each ear at the shen men point.
  Interventions: Other: Acupuncture
- No Acupuncture (Standard of Care) (No Intervention): If needed, the patient will receive a standard does of oral midazolam (0.5 mg /kg or less, up to 15mg) plus acetaminophen 12.5 mg/kg (V group). If the patient does not require premedication with midazolam, oral acetaminophen 12.5mg/kg will be given alone (NV group).
  Induction of anesthesia by mask ventilation with sevoflurane in 50% nitrous oxide mixed with 50% oxygen. Sevoflurane will be incrementally titrated from 0% up to 8%. Nitrous oxide will be discontinued after induction. Anesthesia will be maintained with sevoflurane in an oxygen/air mixture. Sevoflurane concentration will be titrated to maintain the adequate depth of anesthesia. Prior to leaving the operating room, a dose of ketorolac 0.5mg/kg will be given intramuscularly.

INTERVENTIONS:
Other: Acupuncture — If the child is to receive acupuncture, the sites will be cleaned with an alcohol wipe and acupuncture will be performed using a Seirin pionex press needles. A needle will be placed in the Shen Men points of each ear. Needles will also be placed at the left and right Heart 7 (HT-7) point. This acupuncture point is located on the ulnar side of the anterior carpal region, on the palmer crease of the wrist and radial to pisiform bone. The needles will be inserted bilaterally to a depth of 1.8 mm. Needles will not be inserted at a site of active infection or skin breakdown. Needles will remain for the duration of the operation. The needles will be removed before leaving the operating room.
  Arms: Acupuncture

SUMMARY:
Myringotomy tube placement is one of the most commonly performed operations in children. Emergence delirium after such procedures is common. During emergence delirium children can become both a danger to themselves and others around them, including family members and hospital staff.

The primary objective of this study is to determine if acupuncture, when used in combination with standard anesthetic management, decreases the incidence of emergence delirium in pediatric patients following myringotomy tube placement. Patients with and without premedication of midazolam will be included. A secondary objective of this study is to determine our institution's actual incidence of emergence delirium for this operation using a validated scale, the Pediatric Anesthesia Emergence Delirium (PAED) scale. We will also compare rates of emergence delirium in patients that received a premedication of midazolam versus (V) those that did not (NV).

This is a randomized double-blinded trial. We will enroll 100 children aged 1-6 years old. Premedication with midazolam will be decided by the anesthesiologist. If needed, the patient will receive a standard does of oral midazolam plus acetaminophen (V). If the patient does not require premedication with midazolam, oral acetaminophen will be given alone (NV).

Patients will then be randomized to receive either acupuncture with standard general anesthesia care (A) or to receive standard anesthetic care alone (S). Patients, their family members and recovery registered nurses (RNs) will not know if acupuncture was performed. Intraoperative anesthetic techniques will be standardized and include inhaled inductions with nitrous oxide and sevoflurane. Anesthesia maintenance will be inhaled sevoflurane and the usual pain medication ketorolac will be given intramuscularly prior to emergence. Acupuncture needles will be placed after anesthesia induction and removed prior to leaving the operating room. A total of 4 needles will be placed, one in each wrist at the Heart 7 (HT7) point and one in each ear at the Shen Men point. The needles will be inserted bilaterally to a depth of 1.8 mm.

In the PACU, a blinded study observer will evaluate the patient at four time points using the PAED scale: time of awakening and 5, 10 & 15 minutes after awakening. Follow up phone calls will be made one day and one week after surgery. Families will be asked about behavior after discharge, sleep and bed-wetting.

DETAILED DESCRIPTION:
Myringotomy tube placement is one of the most commonly performed operations in children, with almost 700,000 completed in the United States each year 1. Common anesthetic management of these cases includes inhalational anesthesia and no intravenous line placement. Sevoflurane is the inhalational agent used most commonly for induction and maintenance of these patients. Emergence delirium after sevoflurane maintenance is common. In a study of children receiving sevoflurane-based anesthetic for MRIs, 47.6% of participants had emergence agitation 2. In a comparison of different emergence delirium scales, Bajwa and colleagues detected emergence delirium in 32% of subjects using the Pediatric Anesthesia Emergence Delirium (PAED) scale 3. Emergence delirium can be distressing for both children and their caregivers. During emergence delirium children can become both a danger to themselves and others around them, including family members and hospital staff. Emergence delirium can also delay discharge from the post-operative care unit (PACU).

There has been some published evidence that intraoperative acupuncture can decrease the incidence of post-operative delirium. One study enrolled 60 children undergoing bilateral ear tube placement and randomized half of the patients to receive acupuncture at points LI-4 (he gu) and HT-7 (shen men). The acupuncture group had a lower incidence of emergence agitation than the control group at time of arrival in the PACU and during the following 30 minutes 4. This study did not include patients that had received pre-medication with midazolam. It also did not use a validated assessment for emergence delirium in children.

A small retrospective review of 12 children that received acupuncture found that 83% did not show signs of emergence delirium. These patients had needling at 3 locations (SP 6, HT 7, Liv 3) and magnets placed at the ear shen men area. The anesthetic technique used for these patients was not standardized and there was no comparison group.

The primary objective of this study is to determine if acupuncture, when used in combination with standard anesthetic management, decreases the incidence of emergence delirium in pediatric patients following myringotomy tube placement. Patients with and without premedication of midazolam will be included as it is common that children receive sedating medications to facilitate separation from their caregivers.

A secondary objective of this study is to determine our institution's actual incidence of emergence delirium after this operation. We can also compare rates of emergence delirium with or without premedication of midazolam. Emergence delirium will be evaluated using a validated pediatric delirium scale. The Pediatric Anesthesia Emergence Delirium (PAED) scale has been tested for reliability and validity in 50 children 5.

Study Design We plan to explore this question with a randomized double blinded trial of acupuncture in children who are undergoing myringotomy tube placement. Patients will be randomized to receive either acupuncture immediately after anesthesia induction (A) or to receive standard anesthetic care only (S). Patients, their family members and recovery registered nurses (RNs) will not know if acupuncture was performed. The researchers observing the patients in the PACU will also be blinded to whether or not the subject received acupuncture. Intraoperative anesthetic techniques will be standardized, including administering the usual pain medication of ketorolac 0.5mg/kg given intramuscularly to each patient prior to emergence. Needles will be placed after anesthesia induction and removed prior to leaving the operating room. A total of 4 needles will be placed, one in each wrist at the HT7 point and one in each ear at the shen men point. Emergence delirium will be assessed with the Pediatric Anesthesia Emergence Delirium (PAED) scale. A follow up phone call will be made on the first post-operative day (POD #1). We will assess continued emergence delirium after discharge from the PACU, as well as a brief assessment on sleeping patterns the night after surgery. A second follow-up phone call will be made one week after surgery. During that call, we will ask about the child's behavior and sleep patterns since the time of surgery.

We do not know our institution's actual incidence of emergence delirium for this operation. We will assume it to be 25% as suggested by the literature. We do not know the effects of pre-medication with midazolam on the incidence of emergence delirium. We will assume a standard deviation of 4, a value consistent with the current published literature. By enrolling 100 subjects we can detect a difference of scores of at least 2.5 points. This enrollment will give us 80% power with an alpha of 0.05. Since the distribution of scores won't be normal, this enrollment target also includes a 15% increase to allow for a non-parametric distribution of results. Group (A) and group (S) will each have 50 children.

ELIGIBILITY:
Inclusion Criteria:

* children ages 1 - 6 years old with ASA physical status of 1-3
* scheduled for unilateral or bilateral myringotomy tube placement only.

Exclusion Criteria:

* use of mood altering medications, including anti-epileptic medications.
* genetic abnormalities, including Trisomy 21 (Down syndrome).
* children scheduled for additional surgical procedures to be done in conjunction with myringotomy tube placement.
* Patients scheduled for an overnight admission post operatively.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium (PAED) Score | 0-15 minutes after awakening from general anesthesia in the recovery room
  The start of awakening will be indicated by the time point of first observed, sustained eye opening. In the Post-Anesthesia Care Unit (PACU) and Day Stay units, an observer will evaluate the patient at four time points: time of awakening, 5 minutes after awakening, 10 minutes after awakening and 15 minutes after awakening. The observer will use the Pediatric Anesthesia Emergence Delirium (PAED) evaluation tool evaluate each child for emergence delirium.

SECONDARY OUTCOMES:
Behavior Disturbances on Post-Operative Day 1 (POD1) | 24 hours
  A phone call using a telephone script will be made the following day to ask about the patient's recovery including continued emergence delirium after discharge from the PACU. We will also ask about bed wetting.
Behavior Disturbances one week after surgery (POD 7) | 7 days
  A second follow-up phone call will be made one week after surgery. We will ask questions about the child's behavior, bed wetting and sleep patterns since the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christine S Martin, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University (OHSU), Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Dongen TM, van der Heijden GJ, Freling HG, Venekamp RP, Schilder AG. Parent-reported otorrhea in children with tympanostomy tubes: incidence and predictors. PLoS One. 2013 Jul 12;8(7):e69062. doi: 10.1371/journal.pone.0069062. Print 2013. PMID 23874870
- [Result] Isik B, Arslan M, Tunga AD, Kurtipek O. Dexmedetomidine decreases emergence agitation in pediatric patients after sevoflurane anesthesia without surgery. Paediatr Anaesth. 2006 Jul;16(7):748-53. doi: 10.1111/j.1460-9592.2006.01845.x. PMID 16879517
- [Result] Bajwa SA, Costi D, Cyna AM. A comparison of emergence delirium scales following general anesthesia in children. Paediatr Anaesth. 2010 Aug;20(8):704-11. doi: 10.1111/j.1460-9592.2010.03328.x. PMID 20497353
- [Result] Lin YC, Tassone RF, Jahng S, Rahbar R, Holzman RS, Zurakowski D, Sethna NF. Acupuncture management of pain and emergence agitation in children after bilateral myringotomy and tympanostomy tube insertion. Paediatr Anaesth. 2009 Nov;19(11):1096-101. doi: 10.1111/j.1460-9592.2009.03129.x. Epub 2009 Aug 26. PMID 19709377
- [Result] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210